CLINICAL TRIAL: NCT01525940
Title: PillCam Colon Capsule and CT-colonography in the Evaluation of Patients With Incomplete Conventional Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Guido Costamagna, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCE-CTC
Record Dates: First submitted 2012-01-25; First posted 2012-02-03 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Cancer
Keywords: colon capsule endoscopy; CT-colonography; Patients; incomplete colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colon capsule and CT-colonography (Other): PillCam Colon Capsule Endoscopy (Given® Diagnostic System) ingestion first and CT-colonography about 10-12 hours post-ingestion
  Interventions: Device: PillCam Colon Capsule Endoscopy (Given® Diagnostic System)

INTERVENTIONS:
Device: PillCam Colon Capsule Endoscopy (Given® Diagnostic System) — 2nd-generation CCE is 11.6x31.5 mm size, slightly bigger than previous capsule. It has 2 images with an angle of view increased to 172° degrees for each image. CCE-2 captures 35 images/sec. when in motion and 4 images/sec. when virtually stationary. Capsule battery life is at least 10 hours. The Recorder is an external receiving/recording and transmitting unit that receives data transmitted by the capsule. The portable Recorder consists of an antenna array which attaches to the body, a receiver and memory for accumulation of data during the exam. Data transmission is done via high capacity digital link. Workstation is a modified standard personal computer for reviewing videos generated from images acquired by the capsule, interpretation, analysis of acquired data and generating reports.

SUMMARY:
Colorectal cancer (CRC) is the second most common cause of cancer-related death in the Western world, with 500000 deaths per year worldwide. Colonoscopy is accepted as a primary CRC screening tool in many countries. As a preventative procedure, its main purpose is to enable the early diagnosis of CRC at a curable stage and to identify and remove pre-malignant adenomas. Cecal intubation is associated with an increased detection rate of advanced neoplasia, as 33-50% of advanced neoplasia is located in the proximal colon. Complete colonic evaluation is therefore a well-recognized measure of colonoscopy quality control. Cecal intubation rates of ≥ 90% of all colonoscopies in routine clinical practice and ≥ 95% in screening colonoscopies are recommended. Unfortunately, the cecal intubation rate in daily clinical practice is often lower than the target of ≥ 90%, with reported percentages varying from 76.9% to 98.4%. This means that after an incomplete colonoscopy, malignant and pre-malignant lesions may be missed if further investigation is not pursued. Several explanatory factors for incomplete colonoscopy have been described. After an incomplete conventional colonoscopy, patients are required to undergo another test to complete the visualization of the colon. Options for incomplete examinations because of anatomic reasons include both radiologic and endoscopic means.

CT Colonography (CTC ) permits to visualise the whole colon, is minimally invasive, does not require sedation and is well accepted by the patient.

The PillCam Colon Capsule Endoscopy (Given® Diagnostic System)offers an alternative approach for endoscopic visualization of the colon in patients with an incomplete conventional colonoscopy. Advantages of the PillCam Colon Capsule Endoscopy (PCCE) include the elimination of the need for sedation, the minimally invasive, painless nature of the exam, no need of X-rays and the ability to pursue normal daily activities immediately following the procedure. This is a study that is designed to evaluate the performance of the PCCE in the evaluation of patients with an incomplete colonoscopy, compared to the CT-colonography. PCCE and CT-colonography procedures will be compared in regards to completeness of the procedure and detection of lesions in the colon that would have been missed by the incomplete conventional colonoscopy.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second most common cause of cancer-related death in the Western world, with 500000 deaths per year worldwide. Colonoscopy is accepted as a primary CRC screening tool in many countries. As a preventative procedure, its main purpose is to enable the early diagnosis of CRC at a curable stage and to identify and remove pre-malignant adenomas. Cecal intubation is associated with an increased detection rate of advanced neoplasia, as 33-50% of advanced neoplasia is located in the proximal colon. Complete colonic evaluation is therefore a well-recognized measure of colonoscopy quality control. Cecal intubation rates of ≥ 90% of all colonoscopies in routine clinical practice and ≥ 95% in screening colonoscopies are recommended. Unfortunately, the cecal intubation rate in daily clinical practice is often lower than the target of ≥ 90%, with reported percentages varying from 76.9% to 98.4%. This means that after an incomplete colonoscopy, malignant and pre-malignant lesions may be missed if further investigation is not pursued. Several explanatory factors for incomplete colonoscopy have been described. Patient factors that have been shown to increase the risk of an incomplete examination include advanced age, female sex, previous abdominal/pelvic surgery, and diverticular disease. After an incomplete conventional colonoscopy, patients are required to undergo another test to complete the visualization of the colon. Options for incomplete examinations because of anatomic reasons include both radiologic and endoscopic means.

CT Colonography (CTC ) permits to visualise the whole colon, is minimally invasive, does not require sedation and is well accepted by the patient.

The present role of CTC is the integration as a replacement for barium enema in the case of incomplete colonoscopy. In fact ,since 2006 the American Gastroenterological Association (AGA) Clinical Practice and Economics Committee has endorsed CTC as the method of choice for colon investigation in cases of incomplete colonoscopy and numerous evidence exists in the literature showing a clear superiority of CTC over Barium Enema in the detection of CRC and polyps.

Two large, multicenter trials [the American College of Radiology Imaging Network (ACRIN) trial performed in the USA and Italian Multicenter Polyps Accuracy CTC study (IMPACT)trial testing the performance of CTC in comparison with conventional colonoscopy reported that a negative predictive values in both trials for CTC approaching 100%; this is extremely important in order to reassure negative patients about the significance of the examination.The PillCam Colon Capsule Endoscopy (Given® Diagnostic System)offers an alternative approach for endoscopic visualization of the colon in patients with an incomplete conventional colonoscopy. Advantages of the PillCam Colon Capsule Endoscopy (PCCE) include the elimination of the need for sedation, the minimally invasive, painless nature of the exam, no need of X-rays and the ability to pursue normal daily activities immediately following the procedure. Furthermore, PCCE may be well accepted by the subjects, thereby improving subjects' willingness to undergo a second diagnostic evaluation of the colon after the failure of the first endoscopic examination and comply with colorectal cancer screening recommendations. This is a study that is designed to evaluate the performance of the PCCE in the evaluation of patients with an incomplete colonoscopy, compared to the CT-colonography. PCCE and CT-colonography procedures will be compared in regards to completeness of the procedure and detection of lesions in the colon that would have been missed by the incomplete conventional colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between the ages of 18-75 years.
* Subject is referred for colonoscopy as clinically indicated for any reason. This may include, but not limited to, the investigation of any of the following conditions: rectal bleeding, melena, positive stool testing for occult blood, recent change of bowel habits, screening for colorectal cancer, colonic findings on an imaging study
* Subject in which conventional colonoscopy was incomplete

Exclusion Criteria:

* Subject has dysphagia or any swallowing disorder
* Subject has Congestive heart failure
* Subject has high degree of renal insufficiency
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
* Subject has a cardiac pacemaker or other implanted electromedical device.
* Subject has any allergy or other known contraindication to the medications used in the study
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject with any condition believed to have an increased risk for capsule retention such as Crohn's disease, intestinal tumors, radiation enteritis, or NSAID enteropathy,
* Subject has any condition, which precludes compliance with study and/or device instructions.
* Women who are either pregnant or nursing at the time of screening, who intend to be during the study period, or are of child bearing potential and do not practice medically acceptable methods of contraception
* Subject suffers from life threatening conditions
* Subject currently participating in another clinical study
* Iodine contrast allergy
* Hyperthyroidism
* Inflammatory bowel disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the completeness of colonic exploration in patients with a previous incomplete conventional colonoscopy due to technical failure (not due to inadequate cleansing level). | 12 months

SECONDARY OUTCOMES:
To evaluate the difference in terms of accuracy and completeness between PCCE and CT-colonography | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Guido Costamagna, Professor, Principal Investigator — Catholic University Sacred Heart, Rome Italy
Locations (1):
- Catholic University of Sacred Hearth, Rome, Italy, Italy

REFERENCES:
- [Derived] Spada C, Hassan C, Barbaro B, Iafrate F, Cesaro P, Petruzziello L, Minelli Grazioli L, Senore C, Brizi G, Costamagna I, Alvaro G, Iannitti M, Salsano M, Ciolina M, Laghi A, Bonomo L, Costamagna G. Colon capsule versus CT colonography in patients with incomplete colonoscopy: a prospective, comparative trial. Gut. 2015 Feb;64(2):272-81. doi: 10.1136/gutjnl-2013-306550. Epub 2014 Jun 24. PMID 24964317